CLINICAL TRIAL: NCT05557552
Title: Sequential Chemo-immunotherapy Plus Thoracic Radiotherapy for Elderly And/or Frail Stage III Non-small-cell Lung Cancer Patients Unfit for Concurrent Chemoradiotherapy: an Open Label, Two Cohorts, Prospective Trial
Brief Title: Sequential Chemo-immunotherapy Plus Thoracic Radiotherapy for Elderly And/or Frail Stage III Non-small-cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Shengguang Zhao, Prof., Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021(189)
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-11

CONDITIONS: Non-small Cell Lung Cancer Stage III
Keywords: thoradic radiotherapy; non-small-cell lung cancer; chemo-immunotherapy; survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standar thoracic RT dose (Experimental): Sequential chemo-immunotherapy plus standard dose of thoracic radiotherapy followed by anti-PD-1/PD-L1 maintenance therapy
  Interventions: Radiation: standar thoracic RT dose
- decreased thoracic RT dose (Experimental): Sequential chemo-immunotherapy plus decreased thoracic radiotherapy followed by anti-PD-1/PD-L1 maintenance therapy
  Interventions: Radiation: decreased thoracic RT dose

INTERVENTIONS:
Radiation: standar thoracic RT dose — All the enrolled patients will be patients with NSCLC who did not have PD (determined as per the RECIST v1.1) after 4-6 cycle of platinum-based chemotherapy in combination with an anti-PD-1/L1. Then, those enrolled patients would be treated with standard dose thoracic radiotherapy of 60 Gy/30Fx concurrently with PD-1/PD-L1 maintenance therapy, and the total maintenance therapy time should at least more than 6 months.
  Arms: standar thoracic RT dose
Radiation: decreased thoracic RT dose — All the enrolled patients will be patients with NSCLC who did not have PD (determined as per the RECIST v1.1) after 4-6 cycle of platinum-based chemotherapy in combination with an anti-PD-1/L1. Then, those enrolled patients would be treated with decreased thoracic radiotherapy of 50Gy/25Fx concurrently with PD-1/PD-L1 maintenance therapy, and the total maintenance therapy time should at least more than 6 months.
  Arms: decreased thoracic RT dose

SUMMARY:
Concurrent chemoradiotherapy without disease progression followed by consolidation durvalumab is standard of care for unresectable, stage III non-small-cell lung cancer (NSCLC) (the 'PACIFIC regimen'). However, many patients with poor performance status, older age or comorbidities may be ineligible for chemotherapy due to expected high toxicity. The present study aim to investigate the efficacy and toxicities of sequential chemo-immunotherapy plus thoracic radiotherapy for elderly and/or frail stage III NSCLC patients unfit for concurrent chemoradiotherapy, and to identify the optimal thoracic dose for this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at time of study entry
2. Histologically documented diagnosis of unresectable stage III NSCLC;
3. Fully-informed written consent obtained from patients;
4. Unfit for concurrent chemoradiotherapy as determined by the multi-disciplinary team board due to one of the following reasons: (1) ECOG 2; (2)age≥70;(3) ECOG 1 and CCI≥1；
5. Adequate bone marrow, liver and kidney function
6. Life expectancy of at least 3 months
7. At least one measurable (RECIST 1.1), thoracic lesion that can be irradiated
8. Histologic or cytologic confirmation of small cell lung cancer
9. Adequate pulmonary function with FEV1 >1 L or >30 % of predicted value and DLCO >30 % of predicted value

Exclusion Criteria:

1. Previous chemo-, immuno- or radiotherapy for NSCLC
2. Major surgical procedure last 28 days
3. History of allogenic organ transplantation, autoimmune disease, immunodeficiency, hepatitis or HIV
4. Uncontrolled intercurrent illness
5. Other active malignancy
6. Leptomeningeal carcinomatosis
7. Immunosuppressive medication
8. Pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 12 months after last patient entry
  time from treatment start until death or progression of tumor disease within one year

SECONDARY OUTCOMES:
1-year overall survial | 12 months after last patient entry
  time from treatment start until death with in one year
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 within one year | 12 months after last patient entry
  Safety and Tolerability
5-year overall survival | 5-years after last patient entry
  Time from treatment start until death

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai jiaotong univestigy school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No